CLINICAL TRIAL: NCT05675202
Title: Clinical Trial on Absorption, Metabolism and Excretion of [14C] TQ-B3525 in Chinese Adult Male Healthy Subjects - Research on Material Balance and Biotransformation of [14C] TQ-B3525
Brief Title: Material Balance Study of TQ-B3525
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-I-04
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases; Magnetic Resonance Imaging
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — TQ-B3525

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablet (Experimental): 100 µ Ci [14C] TQ-B3525, 20mg, once in total
  Interventions: Drug: TQ-B3525

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 is a new PI3K α/δ Kinase inhibitor

SUMMARY:
A clinical study to investigate the absorption, metabolism and excretion of [14C] TQ-B3525 in Chinese adult male healthy subjects, aiming to quantitatively analyze the total radioactivity in the excreta of male healthy subjects after oral administration of [14C] TQ-B3525, obtain the data of human radioactive excretion rate and main drainage routes, investigate the distribution in whole blood and plasma, the distribution in plasma and the pharmacokinetics of total radioactivity in plasma, and identify the main metabolites, To determine the main biotransformation pathway and obtain the pharmacokinetic parameters of TQ-B3525 and its metabolites in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male;
* Age: 18-45 years old (including boundary value);
* Body weight: Body mass index (BMI) is between 19 and 26 kg/m2 (including the boundary value), and the weight of the subject is not less than 50 kg;
* Sign the informed consent form voluntarily;
* The subjects were able to communicate well with the researchers and complete the trial according to the protocol.

Exclusion Criteria:

* Those with abnormal and clinically significant results from comprehensive physical examination, vital signs, routine laboratory examination (blood routine examination, blood biochemistry, blood coagulation function, urine routine examination, stool routine examination, glycosylated hemoglobin, lipase, amylase), thyroid function, 12 lead ECG, chest CT, abdominal B ultrasound (liver, gallbladder, pancreas, spleen and kidney), etc;
* Abnormal ophthalmic examination (slit lamp, intraocular pressure and fundus photography) with clinical significance;
* Hepatitis B surface antigen or E antigen, anti HCV IgG, HIV Ag/Ab and Treponema pallidum antibody positive;
* Cytomegalovirus (CMV) antibody positive;
* Novel coronavirus nucleic acid positive;
* Any drugs that inhibit or induce liver drug metabolizing enzymes were used within 30 days before the screening period (see Appendix 1 for details);
* Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicine or food supplements, such as vitamins and calcium supplements, within 14 days before the screening period;
* Any serious clinical disease history or any disease or circumstance that the researcher thinks may affect the test results, including but not limited to the history of circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases;
* People with any disease that increases the risk of elevated blood sugar, such as those with a history of primary diabetes, steroid induced diabetes or other secondary diabetes, and those with acute or chronic pancreatitis;
* People who have a history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, history of torsade, ventricular tachycardia, atrioventricular block, history of prolonged QT syndrome, or symptoms of prolonged QT syndrome and family history (certified by genetics or sudden death of a close relative due to cardiac causes when young);
* History of interstitial lung disease, severe impairment of lung function, severe pulmonary fibrosis, radiation pneumonitis, drug-induced lung disease, and chest CT findings during screening period suggest evidence of active pulmonary inflammation;
* Major surgery or incomplete healing of surgical incision within 6 months before the screening period; Major surgery includes, but is not limited to, any surgery with significant bleeding risk, extended general anesthesia period, or open biopsy or obvious traumatic injury;
* Allergic constitution, such as known history of allergy to two or more substances; Or the investigator may be allergic to the test drug or its excipients;
* Hemorrhoids or perianal diseases, irritable bowel syndrome, inflammatory bowel disease with regular/ongoing blood in the stool;
* People with multiple factors affecting oral administration and drug absorption (such as inability to swallow, gastrointestinal resection, ulcerative colitis, symptomatic/inflammatory bowel disease, intestinal obstruction, etc.); habits and customs:
* Habitual constipation or diarrhea;
* Excessive drinking or regular drinking within 6 months before the screening period, that is, drinking more than 14 units of alcohol every week (1 unit=360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine); Or the results of alcohol breath test during screening period ≥ 20 mg/dl;
* Those who smoke more than 5 cigarettes a day or habitually use nicotine containing products in the first 3 months of the screening period and cannot quit during the trial period;
* Abuse of drugs or use of soft drugs (such as marijuana) 3 months before the screening period or use of hard drugs (such as cocaine, amphetamines, and phencyclidine) 1 year before the screening period; Or positive urine drug test during screening period;
* Those who habitually drink grapefruit juice or excessive tea, coffee and/or caffeinated drinks, and cannot give up during the test; other:
* Workers who need to be exposed to radioactive conditions for a long time; Or those who have significant radiation exposure (≥ 2 chest/abdomen CT, or ≥ 3 other kinds of X-ray examinations) or participated in the radiopharmaceutical labeling test within 1 year before the test;
* Those who have a history of needle fainting and blood fainting, and who have difficulty in blood collection or can not tolerate venous puncture blood collection;
* Participated in any other clinical trials (including drug and device clinical trials) within 3 months before the screening period;
* Those who have been vaccinated within one month before screening or who plan to be vaccinated during the trial period;
* hose who have fertility or sperm donation plans during the trial and within one year after the completion of the trial, or those who do not agree that the subject and his/her spouse should take strict contraceptive measures during the trial and within one year after the completion of the trial (see Appendix 3 for details);
* People who have lost blood or donated blood up to 400 mL within 3 months before the screening period, or received blood transfusion within 1 month;
* Subjects who are considered by the researcher to have any factors unsuitable for this experiment.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult male
Enrollment: 8 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Before administration, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after administration
  Maximum plasma drug concentration
Area under drug time curve (AUC 0-t) | Before administration, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after administration
  Area under the plasma concentration time curve from time 0 to last time of quantifiable concentration
Area under drug time curve (AUC 0-last) | Before administration, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after administration
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite time

SECONDARY OUTCOMES:
Incidence rate of adverse events | Before the first administration until it returns to normal or the level considered acceptable by the investigator
  Record the number of cases, time of adverse events, including the abnormal changes in in physical examination, vital signs, 12 lead ECG, laboratory test values and other indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China